CLINICAL TRIAL: NCT05095701
Title: An Open Clinical Trial to Evaluate the Immunity Persistence of Live Attenuated Varicella Vaccine At 5 and 8 Years After Primary Immunization with Live Attenuated Varicella Vaccine
Brief Title: An Immunity Persistence Study of Live Attenuated Varicella Vaccine
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-VZV-4004
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): 349 subjects who enrolled in the experimental group of clinical trial and included in the immunogenicity subgroup PPS set from August to September 2016 will be collected venous blood 3.0~3.5ml at 5 and 8 years after primary immunization.
  Interventions: Biological: Investigational Live Attenuated Varicella Vaccine
- Control Group (Placebo Comparator): 354 subjects who enrolled in the control group of clinical trial and included in the immunogenicity subgroup PPS set from August to September 2016 will be collected venous blood 3.0~3.5ml at 5 and 8 years after primary immunization.
  Interventions: Biological: Placebo (Freeze Dired Dilution)

INTERVENTIONS:
Biological: Investigational Live Attenuated Varicella Vaccine — The live attenuated varicella vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. Live attenuated varicella-virus in 0·5 mL injection water with sucrose,sodium glutamate,sodium chloride,potassium chloride, sodium dihydrogen phosphate, potassium dihydrogen phosphate per injection.
  Arms: Experimental Group
Biological: Placebo (Freeze Dired Dilution) — The placebo (freeze dired dilution) was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. and contained no active ingredient.It was 0·5 mL injection water with sucrose,sodium glutamate,sodium chloride,potassium chloride and phosphate.
  Arms: Control Group

SUMMARY:
This an open phase Ⅳ clinical trial of live attenuated varicella vaccines manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd .The purpose of this study is to evaluate the immunity persistence of live attenuated varicella vaccine at 5 and 8 years after primary immunization with live attenuated varicella vaccine.

DETAILED DESCRIPTION:
This study is an open phase Ⅳ clinical trial in subjects who enrolled in the clinical trial and included in the immunogenicity subgroup PPS set from August to September 2016 .The experimental vaccine and placebo (Freeze Dired Dilution) were manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.A total of 703 subjects will be enrolled including 349 subjects in experimental group and 354 subjects in control group .And 3.0-3.5ml of venous blood was collected from all subjects at 5 and 8 years after primary immunization, and the serum was separated for varicella antibody detection. The window period of blood collection was six months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in PPS immunogenicity subgroup of phase Ⅲ clinical trial of protective effect of varicella vaccine;
* The subject and/or guardian can understand and voluntarily sign the informed consent form;
* Proven legal identity.

Exclusion Criteria:

* History of chickenpox or shingles;
* History of varicella vaccination since phase Ⅲ clinical trial;
* Autoimmune disease or immunodeficiency / immunosuppression;
* History of immunosuppressive therapy since phase Ⅲ clinical trial;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 703 (Estimated)
Dates: Start 2021-12-18 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-seropositive rates of varicella antibody | 5 years after primary immunization
  The seropositive rates of varicella antibody in 5 years after primary immunization with varicella vaccine
Immunogenicity index-GMT of varicella antibody | 5 years after primary immunization
  GMT of varicella antibody in 5 years after primary immunization with varicella vaccine
Immunogenicity index-the seropositive rates of varicella antibody | 8 years after primary immunization
  The seropositive rates of varicella antibody in 8 years after primary immunization with varicella vaccine
Immunogenicity index-the GMT of varicella antibody | 8 years after primary immunization
  GMT of varicella antibody in 8 years after primary immunization with varicella

CONTACTS AND LOCATIONS:
Overall Officials: Lili Huang, Bachelor, Principal Investigator — Henan Provincial Center for Disease Prevention and Control
Locations (2):
- China (2):
  - Xiangcheng County Center for Disease Control and Prevention, Xuchang, Henan
  - Biyang County Center for Disease Control and Prevention, Zhumadian, Henan